CLINICAL TRIAL: NCT05535140
Title: Chatbot Powered G8 Screening Intervention
Brief Title: A Chatbot-Powered G8 Screening Intervention to Facilitate Referrals to a Comprehensive Geriatric Assessment Among Older Adults With Cancer
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kuang-Yi Wen, Associate Professor - Medical Oncology, Thomas Jefferson University
Other Study IDs: 21F.675; 080-27000-S45501 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2022-06-17; First posted 2022-09-10 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Geriatric Cancer Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer patients who are 65 years of age or older: An online self-reported G8 screening tool. The tool will have content including: 1) the purpose and benefit of the G8, 2) explanations of each question with examples and probes to help with recall, and 3) next steps after the G8 assessment is completed and how the results might impact their cancer treatments. New established older cancer patients will be invited to interact with the tool.
  Interventions: Other: G8 Screening Tool

INTERVENTIONS:
Other: G8 Screening Tool — Determine the feasibility of implementing an online patient self-reported G8 assessment, on new patients >65y/o who are scheduled with the medical oncology department.

SUMMARY:
In this prospective quality improvement study, we will develop and evaluate the feasibility and acceptability of an online patient self-reported G8 screening tool which will allow us to efficiently identify G8 positive older cancer patients to be referred to our Senior Adult Oncology Center (SAOC) for a Comprehensive Geriatric Assessment (CGA).

DETAILED DESCRIPTION:
We will test the feasibility and acceptability of the online G8 screening tool developed. 100 older new established cancer patients who had used the MyChart G8 will be recruited to provide their feedback on the usability of the screening tool and any related referral and SAOC appointment experience. Among patients with G8 scores ≤ 14, they will be referred to a CGA. We will examine CGA attendance compliance, predictive value of the online collected G8 score with the final frailty designation determined by the CGA, and perceived barriers among CGA non-adherent patients via a brief follow up inquiry.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older
* New Patient Visit scheduled for Medical Oncology

Exclusion Criteria:

• Inability to answer or have caregiver answer questions on screening tool.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Cancer patients who are 65 years of age or older coming to the medical oncology department at Thomas Jefferson University for care.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Agree to using the G8 assessment | At time of visit
  To determine the feasibility of implementing an online patient self-reported G8 assessment, on new patients >65y/o who are scheduled with the medical oncology department.
Complete the G8 assessment | At time of visit
  To determine the feasibility of implementing an online patient self-reported G8 assessment, on new patients >65y/o who are scheduled with the medical oncology department.
3. Complete the referred SAOC visits if they complete the G8 assessment and are screened positive | After visit
  To determine the feasibility of implementing an online patient self-reported G8 assessment, on new patients >65y/o who are scheduled with the medical oncology department.

CONTACTS AND LOCATIONS:
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States